CLINICAL TRIAL: NCT05138042
Title: Effect of Cryotherapy on Paclitaxel-Induced Peripheral Neuropathy of the Hand in Female Breast Cancer Patients: A Prospective Self-Controlled Study
Brief Title: Chemotherapy - Induced Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, Hsiang Chu Pai, Principal Investigator, Chung Shan Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CS2-19004
Record Dates: First submitted 2021-11-01; First posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Breast Cancer Female
Keywords: peripheral neuropathy; cryotherapy; frozen gloves
MeSH Terms: conditions — Peripheral Nervous System Diseases | interventions — Cryotherapy

STUDY DESIGN:
Intervention Model Description: Frozen glove was provided for dominant hand of breast cancer patients while receiving paclitaxel treat, and as the experimental group. In addition, another hand as a control group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention side (Experimental): Breast cancer patients wore frozen glove on the dominant hand for 90 minutes during their weekly treatment with paclitaxel (80 mg/m2). Treatment was continued for 12 weeks, with their non-dominant hand as the control side
  Interventions: Other: Cryotherapy (frozen glove)
- Control side (No Intervention): Breast cancer patients wore frozen glove on the dominant hand for 90 minutes during their weekly treatment with paclitaxel (80 mg/m2). Treatment was continued for 12 weeks, with their non-dominant hand as the control side

INTERVENTIONS:
Other: Cryotherapy (frozen glove) — In this study, the cryotherapy interventions were based on previous studies, with the dominant hand wearing the frozen glove set as the experimental group, and the non-dominant hand that was not wearing a frozen glove as the control group.
  The cold temperature of the refrigerator was measured in advance to be -20.2°C to -22.8°C. The freezing of the gloves lasted for at least three hours, and the gloves were tested with an infrared temperature-measuring instrument before use. Its temperature range was -24.3°C to -24.7°C. The patient began to wear gloves 15 minutes before the administration of paclitaxel for one hour, and replaced them with new frozen gloves at the 45th minute. The patient continued to wear the gloves until 15 minutes after the end of the chemotherapy drug administration, for a total of 90 minutes.
  Arms: Intervention side

SUMMARY:
The purpose of this study was to examine the efficacy of cryotherapy with frozen gloves for the prevention of the chemotherapy-induced peripheral neuropathy (CIPN) of the hand.

Frozen glove was provided for dominant hand of breast cancer patients while receiving paclitaxel treat, and as the experimental group. In addition, another hand as a control group. The questionnaire was used before chemotherapy and at the fourth, eighth, twelfth, and sixteenth weeks to understand the effectiveness of frozen gloves.

DETAILED DESCRIPTION:
In this study, the cryotherapy interventions were based on previous studies, with the dominant hand wearing the frozen glove set as the experimental group, and the non-dominant hand that was not wearing a frozen glove as the control group. The Elasto-Gel flexible frozen glove (Southwest Technologies, North Kansas City, MO, USA) used in this study lasted for 20 to 40 minutes and was easy to clean.The cold temperature of the refrigerator was measured in advance to be -20.2°C to -22.8°C. The freezing of the gloves lasted for at least three hours, and the gloves were tested with an infrared temperature-measuring instrument before use.

Its temperature range was -24.3°C to -24.7°C. The patient began to wear gloves 15 minutes before the administration of paclitaxel for one hour, and replaced them with new frozen gloves at the 45th minute. The patient continued to wear the gloves until 15 minutes after the end of the chemotherapy drug administration, for a total of 90 minutes. These intervention procedures were used for each treatment for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Women with breast cancer diagnosis confirmed by a physician and receiving paclitaxel for the first time.
* Above 20 years of age.

Exclusion Criteria:

* Patients with neurological disease histories.
* Patients with histories of the hand-foot syndrome.
* Patients with distant cancer metastases or skin metastases.
* Patients with nail lesions or the absence of fingers.
* Patients with a low tolerance to cold, and edema.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-10-07 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
peripheral neuropath (hand sensory symptoms and hand motor symptoms) "change" is being assessed. | Questionnaire were filled out five times, before the first chemotherapy session and at the fourth, eighth, twelfth, and sixteenth weeks following the first chemotherapy session.
  The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Chemotherapy-Induced Peripheral Neuropathy 20 (EORTC QLQ-CIPN 20) was used to assess chemotherapy-induced peripheral neuropathy in breast cancer patients. It contains 20 items and includes three scales (sensory scale, motor scale, and autonomic scale)
  In this study, we focused on the evaluation of the peripheral neurological symptoms of the hand according to the purpose of the research. Therefore, we selected the scope related to the hand in the EORTC QLQ-CIPN20 as an assessment item. It contains four items about sensory symptoms and four items about motor symptoms.Each item is rated on a 4-point Likert-type scale ranging from 1 (not at all) to 4 (very much). The total score is the sum of all item scores. Higher scores reflect more peripheral neuropathic signs and symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Chung Shan Medical University, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No
We have no plan to provide IPD.